CLINICAL TRIAL: NCT02302495
Title: A Multicenter Open Label Phase 2 Study of Carfilzomib Weekly Plus Melphalan and Prednisone in Untreated Symptomatic Elderly Multiple Myeloma
Brief Title: Study of Carfilzomib Weekly Plus Melphalan and Prednisone in Untreated Symptomatic Elderly Multiple Myeloma
Acronym: IFM2012-03
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012_32; 2012-004490-10 (EudraCT Number)
Record Dates: First submitted 2014-11-12; First posted 2014-11-27 (Estimated); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma
Keywords: Carfilzomib weekly; and Melphalan and Prednisone
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; Melphalan; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Carfilzomib weekly+Melphalan+Prednisone (Other): one arm, two steps and two parts.In the first step of the study: 5 cohorts of 6 patients with Carfilzomib weekly administrated at different dose regimen will be opened one after the other to determine Maximum tolerated dose of Carfilzomib based on definition of Dose-limiting toxicities.In the second step of the study:expanded Cohort, 50 patients received Carfilzomib at the MTD. In Part 1. Induction.Nine 5 weeks cycles of weekly CMP are plannedCarfilzomib. 36, 45, 56 or 70 mg/m² on days 1, 8, 15, 22 IV route . Patients will start the first cycle day 1 with 20mg/m². In combination with oral Melphalan 0.25mg/kg/j and oral prednisone 60mg/m², both on days 1 to 4.Part 2. Maintenance.Carfilzomib. 36 mg/m² weekly, every two weeks IV route for 1 year.
  Interventions: Drug: Carfilzomib

INTERVENTIONS:
Drug: Carfilzomib — DOSING REGIMEN.
  The regimen will have 2 parts:
  Part 1. Induction. Nine 5 weeks cycles (35-days each) of weekly Carfilzomib Melphalan Prednisone are planned Carfilzomib. 36, 45, 56 or 70 mg/m² on days 1, 8, 15, 22 IV route followed by a 13-day rest period per 35-days cycle. Patients will start the first cycle day 1 with 20mg/m².
  In combination with oral Melphalan 0.25mg/kg/j and oral prednisone 60mg/m², both on days 1 to 4.
  Part 2. Maintenance. Carfilzomib. 36 mg/m² weekly, every two weeks IV route for 1 year. Melphalan and Prednisone is not pursued at this phase of the study.
  Other Names: Melphalan; Prednisone

SUMMARY:
IFM 2012-03 protocol is a Phase 2 multicenter nonrandomized open in elderly patients with multiple myeloma at diagnosis. Study primary objectives are in the first step to determine Maximum tolerated dose (MTD) of Carfilzomib Weekly based on definition of Dose-limiting toxicities (DLTs) and in the second step to expanded cohort, to determine the VGPR (Very Good Partial Response) + CR (Complete Response) rate of Carfilzomib Weekly at the MTD in combination with Melphalan Prednisone at the end of the 9 induction cycles.

DETAILED DESCRIPTION:
Overall design. This study is a Multicenter, Open-label, Phase 2 study of Carfilzomib Weekly +MP in Untreated Elderly MM. Eligible patients must have a symptomatic, untreated MM with a measurable disease. There is a dose escalation part in the study as the MTD remained to be determined for carfilzomib weekly given for 4 infusions (day 1, 8, 15, 22) on a 35-days cycle.

This study will thus comprise 2 parts. Step 1. To determine MTD of Carfilzomib Weekly based on definition of DLTs - (N=6 patients per cohort, maximum 5 cohorts of carfilzomib weekly +MP) The patients will be included into three cohorts at 36 mg/m², 45 mg/m², 56 mg/m² and 70mg/m² of Carfilzomib Weekly given for 4 infusions (day 1, 8, 15, 22) +MP given on days 1 to 4 of a 35-days cycle. Carfilzomib will be administered at a dose of 36mg/m² for the first cohort where the 20 mg/m² dose is administered on Day 1 of Cycle 1 only and then 36 mg/m² for all subsequent doses.

If dose-limiting toxicities (DLTs) occur in fewer or equal than 2 of these patients, the next cohort of 6 patients (cohort 2) will be opened and patients will receive a dose of 20/45 mg/m². If DLTs occur in fewer or equal than 2 of the patients in cohort 2, the third cohort of 6 patients will receive a dose of 20/56 mg/m² where the 20 mg/m² dose is administered on Day 1 of Cycle 1 only and then 56 mg/m² for all subsequent doses. If DLTs occur in fewer or equal than 2 of the patients in cohort 3, the fourth and five cohort of 6 patients will receive a dose of 20/70 mg/m² where the 20 mg/m² dose is administered on Day 1 of Cycle 1 only and then 70 mg/m² for all subsequent doses.

If at any time during cycle 1 of a dose cohort, > 2 subjects experience a drug-related DLT, the MTD will have been exceeded, additional enrolment within the cohort will cease, and dose escalation will stop. The MTD will be defined as the dose level below which DLT is observed in > 33% (i.e. > 2 of 6) subjects in a cohort.

The following are defined as DLTs:

* Any hematologic toxicity of grade 4 intensity or preventing administration of 2 or more of the 4 carfilzomib doses of the first treatment cycle
* Grade ≥ 3 febrile neutropenia
* Grade ≥ 3 gastrointestinal toxicities
* Any other grade ≥ 3 nonhematologic toxicity considered related to CMP by the principal investigator.
* Grade ≥ 3 peripheral neuropathy persisting for more than 3 weeks after discontinuation of study drugs.

Exceptions are:

1. grade 4 thrombocytopenia without bleeding lasting ≤ 7 days or
2. grade 4 neutropenia lasting ≤ 7 days
3. grade ≥ 3 nausea/ vomiting if the patient had not received adequate antiemetic prophylaxis Adverse events (AEs) will be graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE, version 4.0). MTD determination will be based on occurrence of DLTs during the first induction treatment cycle only.

Step 2. Expanded Cohort (N=50 patients; Carfilzomib weekly at the MTD +MP only) After identification of the MTD, it is planned for the dose cohort to be expanded to include up to a total of 50 patients treated at the MTD of carfilzomib weekly for the step 2 of the study. A full treatment course is the same as for step 1, see "dosing regimen".

ELIGIBILITY:
Inclusion Criteria:

* able to understand and voluntarily sign an informed consent form
* able to adhere to the study visit schedule and other protocol requirements.
* age ≥ 65 years.
* life expectancy > 6 months.Patients must have Symptomatic Measurable previously Untreated MM
* have measurable disease as defined by the following: quantifiable monoclonal M-component value in the serum and/or urine
* eastern Cooperative Oncology Group performance status score ≤2
* dequate bone marrow function, documented within 72 hours and without transfusion 5 days prior to the first intake of investigational product no growth factor support Adequate organ function
* subjects affiliated with an appropriate social security system.
* male subjects must:Understand the potential teratogenic,and genotoxic risk of Melphalan if engaged in sexual activity with a pregnant female or a female of childbearing potential.
* understand the potential genotoxic risk of Carfilzomib if engaged in sexual activity with a pregnant female or a female of childbearing potential.
* practice complete abstinence or understand the need and agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential throughout the entire duration of study treatment, during dose interruptions and until at least 3 months after the end of treatment discontinuation of CMP, even if he has undergone a successful vasectomy.
* if pregnancy or a positive pregnancy test does occur in the partner of a male study patient during study participation, the investigator must be notified immediately.
* agree not to donate semen or sperm during study drug therapy and until at least 3 months after the end of treatment discontinuation of CMP.

Exclusion Criteria:

* any other uncontrolled medical condition or comorbidity that might interfere with subject's participation.
* known positive for HIV or active infectious hepatitis, type B or C.
* patient with terminal renal failure that require dialysis and clearance creatinine < 30 ml/min.
* prior history of malignancies, other than multiple myeloma, unless the patients has been free of the disease for ≥ 5 years.
* prior local irradiation within two weeks before first dose
* evidence of central nervous system (CNS) involvement.
* unable to take corticotherapy at study entry
* any ongoing adverse event or medical history > grade 2 severity
* persons protected by a legal regime (guardianship, trusteeship).Alkeran's (Melphalan) contraindication: Hypersensitivity to Melphalan or to any other constituents.
* patients with heart failure class 3 and 4 according to the NYHA criteria, or patients with past history of myocardial infarction within the last 6 months or no controlled cardiac conduction abnormalities.
* patients with a left ventricular ejection fraction under or equal to 45 % (LVEF ≤ 45%)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-01-08 (Actual); Primary Completion 2016-07-17 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Dose Maximum Tolerate of Carfilzomib Weekly | 35 days
  If dose-limiting toxicities occur in fewer than 3 of these patients per cohort, the next cohort of 6 patients (cohort 2,3 and 4) will be open. If at any time during cycle 1 of a dose cohort, > 2 subjects experience a drug-related dose-limiting toxicities, the Maximum Tolerate Dosing will have been exceeded, additional enrolment within the cohort will cease, and dose escalation will stop. The Maximum Tolerate Dosing will be defined as the dose level below which dose-limiting toxicities is observed in >33% subjects in a cohort.

SECONDARY OUTCOMES:
number of patients who reach Very Good Partial Response and Complete | 315 days
  Expanded cohort, the primary endpoint is the Very Good Partial Response and Complete Response rate of Carfilzomib Weekly at the Maximum Tolerate Dosing and melphalan prednisone at the end of the 9 induction cycles using International Myeloma Working Group response criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Leleu Xavier, MD, PhD, Study Chair — University Hospital
Locations (33):
- France (33):
  - Centre Hospitalier H. Duffaut, Avignon
  - Centre Hospitalier de la côte basque, Bayonne
  - Hôpital Jean Minjoz, Besançon
  - Institut Bergonie, Bordeaux
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Centre Hospitalier William Morey, Chalon-sur-Saône
  - Centre Hospitalier de Chambery, Chambéry
  - Hôpital St Antoine Béclére, Clamart
  - CH Louis Pasteur, Colmar
  - CH Francilien, Corbeil-Essonnes
  - CHU Henri Mondor, Créteil
  - Hématologie Clinique, CHU, Hôpital d'Enfants, Dijon
  - Centre hospitalier départemental La Roche sur Yon, La Roche-sur-Yon
  - Centre Jean Bernard, Le Mans
  - Hôpital St Vincent de Paul - GH-ICL, Lille
  - Chru Lille, Lille
  - CHU de Limoges, Limoges
  - Hématologie, Institut Paoli Calmette, Marseille
  - CH Meaux, Meaux
  - Hôpital Notre Dame de Bon Secours, Metz
  - Hopital J Monod, Montivilliers
  - Hôpital E Muller, Mulhouse
  - CHRU, Hôtel Dieu, Nantes
  - Centre de NICE 2/ Hôpital Archet, Nice
  - CHU Nimes CAREMEAU, Nîmes
  - Hôpital St Antoine, Paris
  - Groupe hospitalier Pitié Salpétrière, Paris
  - Hôpital Haut-Leveque, Pessac
  - Unité de Recherche Clinique - CH Perigueux, Périgueux
  - Centre Hospitalier Lyon Sud -1, Pierre-Bénite
  - Hématologie Clinique, Hôpital Robert Debré, CHU Reims, Reims
  - Hématologie, IUCT oncopole, Toulouse
  - CHRU, Hôpitaux de Brabois, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: Undecided